CLINICAL TRIAL: NCT06581926
Title: A Comparative Analysis of Nutritional Knowledge, Reward-related Eating Behaviours and Body Awareness by Gender in a Cohort of Healthy Young Adults.
Brief Title: A Comparative Analysis of Healthy Young Adults Stratified by Gender.
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Asli Demirtaş, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 2024/07-60
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Healthy Young Adults
Keywords: Healthy; People; Gender; Nutrition; Body awareness
MeSH Terms: conditions — Coitus | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female: Healthy young women aged 18-30 years
  Interventions: Other: Behavioral assessment
- Male: Healthy young men aged 18-30 years
  Interventions: Other: Behavioral assessment

INTERVENTIONS:
Other: Behavioral assessment — nutrition knowledge reward-related eating body awareness

SUMMARY:
This project was planned to examine whether there is a difference between nutrition knowledge level, reward-related eating behaviour and body awareness in healthy young adults according to gender.

DETAILED DESCRIPTION:
Nutritional knowledge is among the factors that affect individuals' eating habits and diet quality. Food consumption is rewarding in itself as it increases energy and eliminates hunger (an unpleasant sensation); however, daily experiences show that people often eat without hunger. Individuals with high body awareness are expected to be aware of the changes occurring in their body and to change these changes. In the project, nutrition knowledge level, reward-related eating behaviour and body awareness will be compared according to gender in healthy young adults, and all these values will be evaluated through scales. The study data will be collected with a single interview by face-to-face interview method. Each participant will be informed about the study and their written and verbal consent will be obtained. The application time of the questionnaires is expected to take approximately 10 minutes for each participant. In case of a difference between genders for the values investigated, it is aimed to develop individuals' awareness of these situations. In addition, the relationship between these situations will also be evaluated. It is aimed to create awareness for the situations that are found to be related.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old

Exclusion Criteria:

* Under 18 years old
* not volunteering

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young individuals
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
nutrition knowledge | Baseline
  Nutritional knowledge level for adults: A 5-point Likert-type scale with a total of 32 propositions was formed. The scores obtained from the evaluation criteria of the nutritional knowledge level scale for adults are evaluated as poor, moderate, good and very good. Participants with a basic nutrition score of less than 45 are considered to have a poor level of knowledge, those with a score between 45 and 55 have a moderate level of knowledge, those with a score between 56 and 65 have a good level of knowledge, and those with a score above 65 have a very good level of knowledge. Participants with a food preference score of less than 30 are considered to have poor knowledge, those with a score of 30-36 are considered to have moderate knowledge, those with a score of 37-42 are considered to have good knowledge, and those with a score of more than 42 are considered to have very good knowledge.
reward-related eating | Baseline
  Reward-Related Eating Scale (RED-13): It is a 5-point Likert-type scale consisting of 13 items in 2017. This scale has three sub-dimensions that assess lack of satiety, preoccupation with food and lack of control over eating. A maximum score of 65 and a minimum score of 13 can be obtained from the Red-13 scale. Higher scores on the Red-13 are associated with greater appetite and craving for sweets.
body awareness | Baseline
  Body Awareness Questionarre (BAQ): It is basically a questionnaire that questions body reactions, the individual's estimates of body processes, the disease process and the sleep-wake cycle. It is a Likert-type questionnaire consisting of 18 items and 4 subgroups. A high score from the questionnaire means a high level of body awareness.
descriptive assessment | Baseline
  In the general information form of the young individuals participating in the study, demographic information (gender, age, height, body weight, body mass index, etc.) was included.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gökçe İnbaşı, MSc., Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Bor, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study data will not be shared with third parties. The informed consent form has been prepared and approved in this way.